CLINICAL TRIAL: NCT03814304
Title: Personalized Brain Activity Modulation to Improve Balance and Cognition in Elderly Fallers
Brief Title: Personalized tDCS in Elderly Fallers Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Brad Manor, Assistant Scientist II; Director, Mobility and Brain Function Lab, Hinda and Arthur Marcus Institute for Aging Research, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AG059089-01
Record Dates: First submitted 2019-01-09; First posted 2019-01-24 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Accidental Falls; Aging

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a single site, sham-controlled, double-blinded, randomized trial of tDCS. Participants will perform baseline functional assessments, as well as a structural MRI of the brain. They will then be assigned to a four-week, 20-session intervention of either personalized tDCS or sham (i.e., control) stimulation, via permuted block randomization stratified by sex to ensure that equal numbers of women, and equal numbers of men, are randomized to each arm.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study personnel administering tDCS and the participants will not be aware of tDCS intervention arm assignment. The investigators will ensure such double-blinding by programming the tDCS software with intervention-specific stimulation codes, as supplied by personnel uninvolved in data collection, prior to study initiation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized tDCS (Experimental): Personalized tDCS: This intervention is designed to facilitate the excitability of the left dlPFC. The direct current delivered by any one electrode will not exceed 2.0 mA; the total amount of current from all electrodes will not exceed 4 mA. Each 20-minute session will begin and end with a 60-second ramp up/down of current amplitude to maximize comfort.
  Interventions: Other: Personalized tDCS
- Active-Sham (Sham Comparator): The investigators will use an active sham in which very low-level currents (0.5 mA total) will be transferred between electrodes in close proximity on the scalp throughout the entire 20-minute session. This intervention will be optimized to each participant to deliver currents designed to not significantly influence their cortical tissue, but still mimic the cutaneous sensations induced by tDCS.
  Interventions: Other: Active-Sham

INTERVENTIONS:
Other: Personalized tDCS — The participant will receive 20, 20-minute sessions of personalized tDCS on Monday-Friday, at approximately the same time of day, over four consecutive weeks.
  Arms: Personalized tDCS
Other: Active-Sham — The participant will receive 20, 20-minute sessions of active-sham stimulation on Monday-Friday, at approximately the same time of day, over four consecutive weeks.
  Arms: Active-Sham

SUMMARY:
The objective of this study is to determine if a four-week, 20-session intervention of personalized transcranial direct current stimulation (tDCS), as compared to sham intervention, improves dual task standing and walking performance (Aim 1), as well as other physical (Aim 2) and cognitive (Aim 3) factors on the causal pathway to falls, in older adults who report two or more falls within the past year and fear of falling again in the future, yet who do not have any acute or over neurological or musculoskeletal condition.

Primary endpoints will include the "dual task" costs to gait speed when walking and postural sway speed when standing, as induced by performing a serial subtraction cognitive task (i.e., [(speeddual task - speedsingle task) / speedsingle task) X 100] (Aim 1), the Short Physical Performance Battery (Aim 2), and the Trail Making Test (Part B minus Part A) (AIM 3). Secondary endpoints will include the dual task cost to serial subtraction performance, additional gait and balance outcomes derived from the dual task paradigm, the Timed Up-and-Go, fear of falling, habitual physical activity, and performance within a battery of neuropsychological tests focused on global cognitive function, attention, verbal fluency and memory.

DETAILED DESCRIPTION:
In older adults, falls are costly, consequential and correlated with both physical and cognitive decline. Most falls occur when standing or walking. Many activities require people to stand or walk while performing tasks like talking or making decisions. Such "dual tasking" interferes with the control of standing and walking. This interference, or "cost," is exaggerated in older adults with previous falls and is predictive of future falls. Neuroimaging evidence indicates that standing and walking,especially when dual tasking, activate distributed brain networks including the left dorsolateral prefrontal cortex (dlPFC)-a brain region sub-serving executive function. Thus, strategies that facilitate activation of the left dlPFC and its connected neural networks hold promise to mitigate dual task costs, improve physical and cognitive function, and ultimately, reduce falls.

Transcranial direct current stimulation (tDCS) provides a noninvasive means of selectively modulating cortical excitability. The investigators have shown in younger and older adults that a 20-minute session of tDCS designed to increase excitability of the left dlPFC reduces dual task costs and improves mobility when tested just after stimulation. The investigators have since completed a pilot, sham-controlled trial of a 2-week, 10-session tDCS intervention targeting the left dlPFC in 20 older adults with slow gait and mild-to-moderate executive dysfunction. The intervention was successfully double-blinded and well-attended. tDCS, compared to sham, reduced dual task costs and induced trends towards improved mobility and executive function over a 2-week follow-up. The investigators thus contend that tDCS targeting the left dlPFC holds promise to improve the control of standing and walking-and ultimately reduce falls-in older adults. Still, the size and duration of tDCS-induced benefits to older adult "fallers" have not been established. Moreover, to date, tDCS delivery has attempted to optimize current flow based on a "typical" brain and has thus not accounted for individual differences in skin, skull, cerebrospinal fluid and brain tissue in the aging brain. Such personalization is now possible with the current flow modeling the investigators propose.

The Overall Aim is to compare, in older adults with previous falls, the effects of a personalized tDCS intervention designed to target the left dlPFC on the dual task costs to standing and walking, and other physical and cognitive factors that are on the causal pathway to falls and important to everyday function. The investigators will conduct a randomized, sham-controlled, double-blinded trial with assessments at baseline and post-intervention (immediate, 3-, 6-month follow-up) in 120 non-demented men and women (60 per arm) aged 60 or older who are at risk of falls and report mobility and balance problems and a fear of falling, yet have no major neural or musculoskeletal disorders that explain their falls. The tDCS intervention will comprise 20, 20-minute sessions of tDCS over a 4-week period.

The investigators hypothesize that, in older adults at risk of falls and over a 6-month follow-up, a personalized tDCS intervention targeting the left dlPFC, as compared to sham, will mitigate dual task costs to the control of standing and walking and enhance other metrics of both physical and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 60 or older
* Self-report of mobility and balance problems
* Self-report of fear of falling defined by a "yes" answer to the yes-or-no question "Is the participant worried about falling in the future?"
* Trail Making Test (TMT) Part B time below 75th percentile of age-and education-based norms
* A score of 10 or below on the Short Physical Performance Battery

Exclusion Criteria:

* Inability to stand or walk unassisted for 60 seconds
* Hospitalization within the past three months due to acute illness, or as the result of a musculoskeletal injury significantly affecting gait or balance
* Any unstable medical condition
* a diagnosis of a gait disorder, Parkinson's disease, Alzheimer's disease or dementia, multiple sclerosis, previous stroke or other neurodegenerative disorder
* Chronic vertigo
* Myocardial infarction within the past 6 months
* Active cancer for which chemo-/radiation therapy is being received
* Psychiatric co-morbidity including major depressive disorder, schizophrenia or psychosis
* Chronic use of any sedating medications (sedatives, anti-psychotics, hypnotics, anti-depressants) or change in medication within the previous month
* Legal blindness
* Contraindications to MRI or tDCS, including reported seizure within the past two years, use of neuro-active drugs, the risk of metal objects anywhere in the body, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp
* A score below 22 on the Telephone Interview of Cognitive Status (TICS)
* Mild or severe dementia defined by a Clinical Dementia Rating (CDR) score of one or greater

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the dual task cost to gait speed | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in the degree to which performing a secondary cognitive task diminishes gait speed.
Change from baseline in the dual task cost to standing postural sway speed | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in the degree to which performing a secondary cognitive task diminishes the control of standing posture.
Change from baseline in Short Physical Performance Battery (SPPB) | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in overall physical function.
Change from baseline in Montreal Cognitive Assessment (MoCA) total score | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This common test will assess the change from baseline in global cognitive function

SECONDARY OUTCOMES:
Change from baseline in the dual task cost to serial subtraction performance | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in the degree to which standing or walking diminishes the ability to perform a cognitive task.
Change from baseline in the dual task cost to stride time variability | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in the degree to which performing a secondary cognitive task diminishes the control of gait.
Change from baseline in dual task cost to walking double support time | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in the degree to which performing a secondary cognitive task diminishes the control of gait.
Change from baseline in the dual task cost to standing postural sway elliptical area | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in the degree to which performing a secondary cognitive task
Change from baseline in Trail Making Test B - A | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in cognitive executive function.
Change from baseline in Timed Up-and-Go (TUG) | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in mobility.
Change from baseline in Falls Efficacy Scale | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in fear of falling. Participants will rate, on a 4-point Likert scale, fear of falling when performing 16 activities. Scores are added up to calculate a total score that ranges from 16 to 64. The cut-point for high fear of falling (FOF) is defined as scores >23 for this 16-item scale.
Change from baseline in 5-day accelerometry-based habitual physical activity | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This metric will assess the change from baseline in the quantity and quality of habitual physical activity.
Change from baseline in Digit Span | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This common test will assess the change from baseline in working memory.
Change from baseline in WAIS-IV Coding Test | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This common test will assess the change from baseline in sustained attention and motor speed.
Change from baseline in Category and Phonemic Fluency Test | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This common test will assess the change from baseline in word retrieval
Change from baseline in Hopkins Verbal Learning Test | 3-day follow-up; 3-month follow-up; 6-month follow-up
  This common test will assess the change from baseline in memory

CONTACTS AND LOCATIONS:
Overall Officials: Brad Manor, PhD, Principal Investigator — Hebrew SeniorLife
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The HSL Institute for Aging Research will promote the development of new research and new investigators by making the data available to outside investigators. The database will include longitudinal demographic, clinical, functional, physiologic, and brain imaging data, from all participants.
  All data will be stripped of primary identifiers and entered into a master database. All data collection procedures, variable definitions and codes, field locations, and frequencies will be documented in a separate file.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will make the data and associated documentation available once summary data are published or otherwise made available, starting six months after publication.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: 1) a commitment to using data only for research purposes and not to identify any particular participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed. The availability of data will be advertised over the Internet through websites maintained by Hebrew SeniorLife and Harvard Medical School.
  All investigators wishing to access the data will submit a brief proposal describing their research project, data needs, regulatory approvals, and mechanisms to assure patient confidentiality. Upon affirmative review by the Principal Investigator and co-investigators of this study, a data-sharing agreement will be signed and the requesting investigators will be given a working data file and appropriate documentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT03814304/Prot_SAP_000.pdf